CLINICAL TRIAL: NCT06023836
Title: Myofascial Pain Syndrome in Plantar Fasciitis; Comparison of Dry Needling and Extracorporeal Shockwave Therapy (ESWT) Effects on Pain and Function
Brief Title: Myofascial Pain Syndrome and Plantar Fasciitis Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Burak Tayyip Dede, Medical Doctor, Istanbul Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07/04/2023; 2011-KAEK-50;89
Record Dates: First submitted 2023-08-26; First posted 2023-09-05 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Plantar Fascitis; Myofascial Pain Syndrome
Keywords: plantar fasciitis; ESWT; dry needling
MeSH Terms: conditions — Myofascial Pain Syndromes; Fasciitis, Plantar | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Participants will be randomly divided into 2 groups and will be treated with ESWT or Dry needling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1: ESWT treatment (Active Comparator): Participants in this group will only receive ESWT treatment
  Interventions: Device: ESWT
- Dry needling (Active Comparator): Participants in this group will only receive Dry needling treatment
  Interventions: Procedure: Dry needling

INTERVENTIONS:
Device: ESWT — Patients in this group received three sessions of ESWT (MASTERPLUS MP 200 ENERGY 2 trademarked ESWT device) at an energy density of 2 bars and a frequency of 2,000 shocks/min at 12 Hz for three weeks, each session once a week. Each of the five most sensitive and painful points was given 400 pulses in the supine position
  Arms: group 1: ESWT treatment
Procedure: Dry needling — Dry needling with Seirin branded 0.6*50 mm acupuncture needles will be performed for 3 sessions with one week intervals for the trigger point detected by manual palpation in the medial gastrocnemius, lateral gastrocnemius, soleus, flexor digitorum brevis, quadratus plantae, abductor hallucis brevis muscles of the patients in the group.
  Arms: Dry needling

SUMMARY:
Patients with plantar fasciitis between the ages of 25-65 years who presented to the Physical Medicine and Rehabilitation clinic with the complaint of heel pain and met the inclusion and exclusion criteria will be included in the study. Demographic data (age, gender, body mass index, symptom duration) will be recorded at the beginning of the study. Then, Foot Functional Index (FFI) and Visual Analog Scale (VAS) scales will be recorded. Participants will be randomly divided into two groups. Group 1 will receive dry needling and Group 2 will receive extracorporeal shock wave therapy (ESWT). Patients in the 1st group will undergo 3 sessions of dry needling with Seirin branded 0.6*50 mm acupuncture needles at one week intervals for the trigger point detected by manual palpation in the medial gastrocnemius, lateral gastrocnemius, soleus, flexor digitorum brevis, quadratus plantae, abductor hallucis brevis muscles. Patients in the 2nd group, Patients in this group received three sessions of ESWT (MASTERPLUS MP 200 ENERGY 2 trademarked ESWT device) at an energy density of 2 bars and a frequency of 2,000 shocks/min at 12 Hz for three weeks, each session once a week. Each of the five most sensitive and painful points was given 400 pulses in the supine position

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 25-65 years with heel pain for more than 6 weeks
* tenderness on palpation in the medial calcaneal region
* aggravation of symptoms while standing and in the first hours of the morning
* who agreed not to receive anti-inflammatory treatment during the study period
* fascia thickness >4mm measured by ultrasound.

Exclusion Criteria:

* Patients diagnosed with rheumatologic diseases
* Those diagnosed with Diabetes Mellitus (DM), those with chronic liver and kidney failure
* Anti-inflammatory-analgesic treatment within the last 1 month
* Diagnosed with inflammatory rheumatic disease
* Those with a history of foot surgery
* Those with mid or hindfoot deformity
* Previous history of central or peripheral nerve damage, lower extremity neuropathy
* Those diagnosed with Diabetes Mellitus
* Those with cognitive impairment
* Unassisted mobilization
* Those with bleeding disorders
* Pregnant women

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
Pain was evaluated with a Visual analog scale (VAS) score. | 5 months
  VAS score ranges from 0 to 10.
  Comparison of the effects of ESWT and dry needling on pain in the management of plantar fasciitis
Function was evaluated with (Foot Functional Index) FFI score. | 5 months
  Comparison of the effects of ESWT and dry needling on function in the management of plantar fasciitis

CONTACTS AND LOCATIONS:
Overall Officials: Burak Tayyip Dede, Principal Investigator — İstanbul Training and Research Hospital
Locations (1):
- Istanbul Training and Resarch Hospital, Istanbul, Turkey (Türkiye)